CLINICAL TRIAL: NCT07282223
Title: Contralateral Adrenal Volume Predicts Duration of Postoperative Steroid Replacement Therapy in Non-ACTH-dependent Hypercortisolism
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUFH-CS-CAV-001
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Cushing's Syndrome; Postoperative; Glucocorticoid; Prediction
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational diagnostic model development — observational diagnostic model development

SUMMARY:
To identify preoperative factors influencing the duration of steroid replacement therapy after adrenalectomy/adrenal-sparing surgery in patients with non-ACTH-dependent hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

* In all, 111 patients (meadian age: 54years; 64.9% female) were included and received postoperative steroid replacement therapy, among whom 65 were diagnosed with subclinical Cushing's syndrome (SCS) and 46 with overt Cushing's syndrome (CS).

Exclusion Criteria:

* none

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In all, 111 patients (meadian age: 54years; 64.9% female) were included and received postoperative steroid replacement therapy, among whom 65 were diagnosed with subclinical Cushing's syndrome (SCS) and 46 with overt Cushing's syndrome (CS).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Tumor volume | from 2017 to 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Peking University First Hospital, Beijing, 100034, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes